CLINICAL TRIAL: NCT02931071
Title: Clinical Phase II Trial to Evaluate Efficacy and Safety of CD34+ Cells Mobilization and Collection After Treatment With Plerixafor and Filgrastim in Patients With Fanconi Anemia for Subsequent Transduction With a Lentiviral Vector Carring FANCA Gene and Reinfusion in the Patient
Brief Title: Clinical Phase II Trial to Evaluate CD34+ Cells Mobilization and Collection in Patients With Fanconi Anemia for Subsequent Transduction With a Lentiviral Vector Carring FANCA Gene. FANCOSTEM-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: CIEMAT (Unknown); CIBERER (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FANCOSTEM-1; 2011-006197-88 (EudraCT Number)
Record Dates: First submitted 2016-09-06; First posted 2016-10-12 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Filgrastim; plerixafor

ARMS (1):
- plerixafor and filgrastim treatment (Experimental): to assess the safety and efficacy of CD34+ cells mobilization with plerixafor and filgrastim
  Interventions: Drug: filgrastim; Drug: plerixafor

INTERVENTIONS:
Drug: filgrastim — G-CSF (12 μg/Kg/12 h) 8 days.
Drug: plerixafor — Plerixafor 0,24 mg/kg/day after the fourth day of G-CSF, and until 5 cells CD34+/μL, max 4 doses of plerixafor

SUMMARY:
Fanconi anemia (FA) is a congenital disease characterized by bone marrow failure and increased incidence of malignant tumors. The Project pursue the optimization of the collection of hematopoietic progenitor cells for later use in another clinical trial entitled "Clinical Trial Phase I/II to evaluate the safety and efficacy of the infusion of autologous CD34+ cells mobilized with mozobil and filgrastim, and transduced with a lentiviral vector carrying the FANCA gene (Orphan Drug) for patients with Fanconi Anemia Subtype A ". The objectives of this study are, therefore, to assess the safety and efficacy of CD34+ cells mobilization with mozobil and filgrastim, which is postulated the most efficient for the collection of CD34+ cells from FA patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 1 year
* diagnosed of Fanconi's anemia confirmed by instability chromosomal test with diepoxy-butane or mitomycin C
* At least one of the following parameters must be higher than these values: Hemoglobin:8,0 g/dL; neutrophils: 750/mm3; platelets: 30.000/mm3
* Lansky index> 60%.
* Left ventricular ejection fraction >50%.
* To grant informed consent in agreement with current law norms
* Women in childbearing age must obtain a negative result in the pregnancy test in serum or urine in the visit of selection and accept the use of suitable contraceptive methods since at least 14 days prior to the first dose of mobilizing treatment until the 14 days following the last

Exclusion Criteria:

* Evidence of myelodysplastic syndromes or leukemia, or cytogenetic abnormalities predicted of these syndromes in bone marrow aspiration. Cytogenetic analyses performed 2 months before starting study are accepted
* Patients with active infection process or any other underlaying severe medical process
* Severe Functional alteration of organs (hepatic, renal, respiratory)(?3), according to National Cancer Institute (NCI CTCAE v3) criteria
* Haematopoietic transplant
* Any disease or concomitant process that is not compatible with the study as per investigator opinion
* Patients not elegible because of an psico-social evaluation
* Patients that received transfusional support during the last 3 months.
* Pregnant or breastfeeding women

Ages: 2 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Toxicity of the mobilization procedure according to National Cancer Institute (CTC NCI, versión 3.0) | after 12 months
  At a year (± 30 days) after the last apheresis, a complete physical examination, blood cell count, basic biochemistry and bone marrow aspirate will be done to the patient in order to control their general health status.

SECONDARY OUTCOMES:
Percentage of patients that reach >5 CD34+ cells/mcl after treatment with filgrastim and plerixafor | after 8 days
  mobilization protocol will be determined by the percentage of patients who achieve peripheral blood counts exceeding 5 CD34+ cells /microliter
Percentage of patients that reach a total CD34+ yield >4x10E6/kg, using the estimated weight of the patient in 5 years | after 8 days
  the CD34+ cell collection protocol will be determined by the percentage of patients who reach at least one million CD34 + cells per kilogram of body weight projected to 5 years after the mobilization process
Percentage of samples in which the recovery of CD34+ cells after the immunomagnetic selection procedure is >50% | after 8 days
  the of CD34+ cell selection process will be determined by the proportion of immunoselected samples where the recovery of CD34 + cells is at least 50%, and where the final percentage of CD34+ cells is at least 50%
Percentage of patients in which the CD34+ cells after the immunomagnetic selection is ³ 4x10E6/kg, using the projected weight at 5 years | after 8 days
  will be determined by the percentage of patients who reach at least one million CD34 + cells per kilo of weight projected to 5 years after the immunomagnetic selection process of all the collected cells

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Díaz de Heredia, MD, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (2):
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Madrid

REFERENCES:
- [Derived] Sevilla J, Navarro S, Rio P, Sanchez-Dominguez R, Zubicaray J, Galvez E, Merino E, Sebastian E, Azqueta C, Casado JA, Segovia JC, Alberquilla O, Bogliolo M, Roman-Rodriguez FJ, Gimenez Y, Larcher L, Salgado R, Pujol RM, Hladun R, Castillo A, Soulier J, Querol S, Fernandez J, Schwartz J, Garcia de Andoin N, Lopez R, Catala A, Surralles J, Diaz-de-Heredia C, Bueren JA. Improved collection of hematopoietic stem cells and progenitors from Fanconi anemia patients for gene therapy purposes. Mol Ther Methods Clin Dev. 2021 Jun 12;22:66-75. doi: 10.1016/j.omtm.2021.06.001. eCollection 2021 Sep 10. PMID 34485595